CLINICAL TRIAL: NCT05599958
Title: Clinical and Genetic Profile of Pediatric Patients With Cystic Fibrosis in Sohag.
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Lamiaa Kamel Morssi, resident doctor, Sohag University
Other Study IDs: Soh-Med-22-10-20
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Cystic Fibrosis
Keywords: sweat chloride test; genetics
MeSH Terms: conditions — Cystic Fibrosis | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood sample for genetic testing for CFTR gene
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: sweat chloride test — assessing chloride (Cl-) concentration in sweat of the patient
Genetic: genetic testing — detection of CFTR mutation

SUMMARY:
Cystic fibrosis (CF) is an autosomal recessive genetic disorder caused by mutations in the gene encoding CF transmembrane conductance regulator (CFTR), which is located at 7q31.2 and encodes 1480 amino acids. CFTR protein is responsible for regulating the transport of electrolytes and chloride across epithelial and mucus-producing cell membranes.

DETAILED DESCRIPTION:
The discovery of the CFTR gene in the late 1980s triggered a surge of basic research that enhanced understanding of the pathophysiology and the genotype-phenotype relationships of this clinically variable disease of cystic fibrosis. More than 2000 variants of CFTR gene have been reported, and they are grouped to six classes depending on the pathophysiology of the CFTR protein ,The most common genetic defect reported in CF is the delta F508 mutation, Moreover, the degree of CF severity depends on the type of mutation, which typically affects the function and quantity of CFTR channels. When the CFTR protein is mutated, chloride ions accumulate in mucus-producing cells, resulting in a thick, sticky mucus that obstructs various pathways and hinders pulmonary, digestive, exocrine and male reproductive functions. Furthermore, mucus buildup increases a patient's susceptibility to airway obstruction, bacterial lung infection, pancreatic insufficiency, malabsorption and infertility. CF is characterized by significant clinical heterogeneity.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 2 days - 18 year.
* patients clinically suspected or diagnosed with cystic fibrosis
* patients diagnosed with cystic fibrosis and attending or referred to the Pediatric pulmonology clinic at Sohag University Hospital.

Exclusion Criteria:

* Patient with cystic fibrosis like symptoms with another confirmed diagnosis ex. primary ciliary dyskinesia

Ages: 2 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric pulmonology clinic
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
number of patients presented with each presenting symptoms and signs . | 6 months
  number of patients with each main presenting symptoms of cystic fibrosis as respiratory distress ,dehydration or others .
number of patients affected with different genetic mutations causing cystic fibrosis. | 6 months
  detecting the different genetic mutations affecting pediatric patients in Sohag

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Riordan JR, Rommens JM, Kerem B, Alon N, Rozmahel R, Grzelczak Z, Zielenski J, Lok S, Plavsic N, Chou JL, et al. Identification of the cystic fibrosis gene: cloning and characterization of complementary DNA. Science. 1989 Sep 8;245(4922):1066-73. doi: 10.1126/science.2475911.
- [Background] Al-Sadeq D, Abunada T, Dalloul R, Fahad S, Taleb S, Aljassim K, Al Hamed FA, Zayed H. Spectrum of mutations of cystic fibrosis in the 22 Arab countries: A systematic review. Respirology. 2019 Feb;24(2):127-136. doi: 10.1111/resp.13437. Epub 2018 Nov 12. PMID 30419605
- [Background] Proesmans M. Best practices in the treatment of early cystic fibrosis lung disease. Ther Adv Respir Dis. 2017 Feb;11(2):97-104. doi: 10.1177/1753465816680573. Epub 2016 Dec 2. PMID 27913761
- [Background] Castellani C, Assael BM. Cystic fibrosis: a clinical view. Cell Mol Life Sci. 2017 Jan;74(1):129-140. doi: 10.1007/s00018-016-2393-9. Epub 2016 Oct 5. PMID 27709245
- [Result] Bell SC, Mall MA, Gutierrez H, Macek M, Madge S, Davies JC, Burgel PR, Tullis E, Castanos C, Castellani C, Byrnes CA, Cathcart F, Chotirmall SH, Cosgriff R, Eichler I, Fajac I, Goss CH, Drevinek P, Farrell PM, Gravelle AM, Havermans T, Mayer-Hamblett N, Kashirskaya N, Kerem E, Mathew JL, McKone EF, Naehrlich L, Nasr SZ, Oates GR, O'Neill C, Pypops U, Raraigh KS, Rowe SM, Southern KW, Sivam S, Stephenson AL, Zampoli M, Ratjen F. The future of cystic fibrosis care: a global perspective. Lancet Respir Med. 2020 Jan;8(1):65-124. doi: 10.1016/S2213-2600(19)30337-6. Epub 2019 Sep 27. PMID 31570318